CLINICAL TRIAL: NCT02873260
Title: A Phase 1 Evaluation of the Safety and Protective Efficacy of a Single Dose of the Live Attenuated Tetravalent Dengue Vaccine TV005 to Protect Against Infection With rDEN3Δ30
Brief Title: Evaluating the Safety and Protective Efficacy of a Single Dose of the Live Attenuated Tetravalent Dengue Vaccine TV005 to Protect Against Infection With rDEN3Δ30
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: CIR 309
Record Dates: First submitted 2016-08-16; First posted 2016-08-19 (Estimated); Last update posted 2018-03-08 (Actual); Status verified 2018-03

CONDITIONS: Dengue
Keywords: Dengue Vaccine
MeSH Terms: conditions — Dengue

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- TetraVax-DV-TV005 + rDEN3Δ30 (Experimental): Participants will receive the TetraVax-DV-TV005 vaccine at Day 0 and the rDEN3Δ30 virus at Day 180.
  Interventions: Biological: TetraVax-DV-TV005; Biological: rDEN3Δ30
- Placebo + rDEN3Δ30 (Placebo Comparator): Participants will receive placebo at Day 0 and the rDEN3Δ30 virus at Day 180.
  Interventions: Biological: rDEN3Δ30; Biological: Placebo

INTERVENTIONS:
Biological: TetraVax-DV-TV005 — TetraVax-DV-TV005 contains 10^3.3 plaque forming units (PFU)/mL of rDEN1Δ30, 10^4.3 PFU/mL of rDEN2/4Δ30(ME), 10^3.3 PFU/mL of rDEN3Δ30/31-7164, and 10^3.3 PFU/mL of rDEN4Δ30. The vaccine is administered in 0.5 mL containing 10^3.0 PFU of each component with the exception of rDEN2/4Δ30 that is given at a dose of 10^4 PFU. TetraVax-DV-TV005 is administered by subcutaneous injection in the deltoid region of the upper arm.
  Other Names: TV005
  Arms: TetraVax-DV-TV005 + rDEN3Δ30
Biological: rDEN3Δ30 — Administered at a dose of 10^4 PFU by subcutaneous injection in the deltoid region of the upper arm.
Biological: Placebo — Administered at a volume of 0.5 mL by subcutaneous injection in the deltoid region of the upper arm.
  Arms: Placebo + rDEN3Δ30

SUMMARY:
This study will evaluate the ability of a single dose of the live attenuated recombinant tetravalent dengue vaccine TetraVax-DV-TV005 (referred to as TV005) to protect against infection with rDEN3Δ30, an attenuated DENV-3, when administered 6 months after the TV005 vaccine.

DETAILED DESCRIPTION:
Dengue infection ranging from mild illness to life-threatening disease is widespread in most tropical and subtropical regions of the world. Infection with any of the four serotypes of dengue virus (DENV-1, DENV-2, DENV-3, and DENV-4) can cause dengue illness. TetraVax-DV-TV005 (referred to as TV005) is a live attenuated recombinant tetravalent dengue virus vaccine developed to protect against all four dengue virus serotypes. This study will evaluate the ability of a single dose of TV005 to protect against infection with rDEN3Δ30, a naturally attenuated DENV-3, given 6 months following vaccination with TV005.

This study will enroll healthy adults with no history of previous flavivirus infection. At Day 0 (study entry), participants will be randomly assigned to receive either the TV005 vaccine or placebo. On Day 180, all participants will receive the rDEN3Δ30 virus. All participants will record their temperature 3 times a day for 16 days after each vaccination. Additional study visits will occur on Days 4, 6, 8, 10, 12, 14, 16, 21, 28, 56, 90, 150, 184, 186, 188, 190, 192, 194, 196, 201, 208, 236, 270, and 360. Study visits will include physical examinations and blood collection.

ELIGIBILITY:
Inclusion Criteria:

* Adult male or female between 18 and 50 years of age, inclusive.
* Good general health as determined by physical examination, laboratory screening, and review of medical history.
* Available for the duration of the study, approximately 26 weeks post-second inoculation.
* Willingness to participate in the study as evidenced by signing the informed consent document.
* Females Only: Female subjects of childbearing potential willing to use effective contraception. Reliable methods of contraception include hormonal birth control, condoms with spermicide, diaphragm with spermicide, surgical sterilization, intrauterine device, and abstinence (greater than or equal to 6 months since last sexual encounter). All female subjects will be considered having child-bearing potential except for those with hysterectomy, tubal ligation, tubal coil (at least 3 months prior to vaccination), or post-menopausal status documented as at least 1 year since last menstrual period.

Exclusion Criteria:

* Females Only: Currently pregnant, as determined by positive β-human choriogonadotropin (HCG) test, breast-feeding.
* Evidence of clinically significant neurologic, cardiac, pulmonary, hepatic, rheumatologic, autoimmune, or renal disease by history, physical examination, and/or laboratory studies.
* Behavioral, cognitive, or psychiatric disease that in the opinion of the investigator affects the ability of the subject to understand and cooperate with the requirements of the study protocol.
* Screening laboratory values of Grade 1 or above for absolute neutrophil count (ANC), alanine aminotransferase (ALT), and serum creatinine, as defined in this protocol.
* Any other condition that in the opinion of the investigator would jeopardize the safety or rights of a subject participating in the trial or would render the subject unable to comply with the protocol.
* Any significant alcohol or drug abuse in the past 12 months that has caused medical, occupational, or family problems, as indicated by subject history.
* History of a severe allergic reaction or anaphylaxis.
* Severe asthma (emergency room visit or hospitalization within the last 6 months).
* HIV infection, by screening and confirmatory assays.
* Hepatitis C virus (HCV) infection, by screening and confirmatory assays.
* Hepatitis B virus (HBV) infection, by hepatitis B surface antigen (HBsAg) screening.
* Any known immunodeficiency syndrome.
* Current use of anticoagulant medications (this does not include anti-platelet medication such as aspirin or non-steroidal anti-inflammatory medications).
* Use of corticosteroids (excluding topical or nasal) or immunosuppressive drugs within 28 days prior to or following vaccination. Immunosuppressive dose of corticosteroids is defined as greater than or equal to 10 mg prednisone equivalent per day for greater than or equal to 14 days.
* Receipt of a live vaccine within 28 days or a killed vaccine within the 14 days prior to vaccination or anticipated receipt of any vaccine during the 28 days following vaccination.
* Asplenia.
* Receipt of blood products within the past 6 months, including transfusions or immunoglobulin or anticipated receipt of any blood products or immunoglobulin during the 28 days following vaccination.
* History or serologic evidence of previous dengue virus infection or other flavivirus infection (e.g., yellow fever virus, St. Louis encephalitis virus, West Nile virus). Subjects will also be screened for Zika virus if they have traveled in the past 18 months to areas of South & Central America that have reported Zika-virus transmission (per Centers for Disease Control and Prevention [CDC] Zika travel information).
* Previous receipt of a flavivirus vaccine (licensed or experimental).
* Anticipated receipt of any investigational agent in the 28 days before or after vaccination.
* Subject has definite plans to travel to a dengue endemic area during the study.
* Refusal to allow storage of specimens for future research.

Inclusion Criteria for Second Vaccine:

* Good general health as determined by physical examination and review of medical history.
* Available for the duration of the study, approximately 26 weeks after the second dose.
* Willingness to participate in the study as evidenced by signing the informed consent document.
* Females Only: Female subjects of childbearing potential willing to use effective contraception for the duration of the trial. Reliable methods of contraception include: hormonal birth control, condoms with spermicide, diaphragm with spermicide, surgical sterilization, intrauterine device, and abstinence (greater than or equal to 6 months since last sexual encounter). All female subjects will be considered having child-bearing potential except for those with hysterectomy, tubal ligation, tubal coil (at least 3 months prior to vaccination), or post-menopausal status documented as at least 1 year since last menstrual period.

Exclusion Criteria for rDEN3Δ30 Administration:

* Anaphylaxis or angioedema following the TV005 administration.
* Females Only: Currently pregnant, as determined by positive β- HCG test, breast-feeding.
* Evidence of clinically significant neurologic, cardiac, pulmonary, hepatic, rheumatologic, autoimmune, or renal disease by history, physical examination, and/or laboratory studies.
* Behavioral, cognitive, or psychiatric disease that in the opinion of the investigator affects the ability of the subject to understand and cooperate with the requirements of the study protocol.
* Any other condition that in the opinion of the investigator would jeopardize the safety or rights of a subject participating in the trial or would render the subject unable to comply with the protocol.
* Any significant alcohol or drug abuse in the past 12 months that has caused medical, occupational, or family problems, as indicated by subject history.
* History of a severe allergic reaction or anaphylaxis.
* Severe asthma (emergency room visit or hospitalization within the last 6 months).
* HIV infection, by screening and confirmatory assays.
* HCV infection, by screening and confirmatory assays.
* HBV infection, by HBsAg screening.
* Any known immunodeficiency syndrome.
* Current use of anticoagulant medications (this does not include anti-platelet medication such as aspirin or non-steroidal anti-inflammatory medications).
* Use of corticosteroids (excluding topical or nasal) or immunosuppressive drugs within 42 days prior to or following vaccination. Immunosuppressive dose of corticosteroids is defined as greater than or equal to 10 mg prednisone equivalent per day for greater than or equal to 14 days.
* Receipt of a live vaccine within 28 days or a killed vaccine within the 14 days prior to vaccination or anticipated receipt of any vaccine during the 28 days following vaccination.
* Asplenia.
* Receipt of blood products within the past 6 months, including transfusions or immunoglobulin or anticipated receipt of any blood products or immunoglobulin during the 28 days following vaccination.
* Anticipated receipt of any other investigational agent in the 28 days before or after vaccination.
* Subject has definite plans to travel to a dengue endemic area during the study.
* Refusal to allow storage of specimens for future research.

Other Treatments and Ongoing Exclusion Criteria:

The following criteria will be reviewed on Study Days 28 and 56 following each vaccination. If any become applicable during the study, the subject will not be included in per-protocol immunogenicity evaluations, as of the exclusionary visit. The subject will, however, be encouraged to remain in the study for safety evaluations until 6 months following the last vaccination (or challenge) received. The subject will have samples obtained at the protocol-defined time-points for immunogenicity and will be included in intention-to-treat immunogenicity analysis.

* Use of any investigational drug or investigational vaccine other than the study vaccine during the 28-day period post-vaccination.
* Chronic administration (greater than or equal to 14 days) of steroids (defined as prednisone equivalent of greater than or equal to 10 mg per day), immunosuppressants, or other immune-modifying drugs initiated during the 28-day period post-vaccination (topical and nasal steroids are allowed).
* Receipt of a licensed vaccine during the 21-day period post vaccination.
* Receipt of immunoglobulins and/or any blood products during the 28-day period post-vaccination.
* Pregnancy -see clarifying language in the protocol. If the pregnancy is terminated spontaneously or by therapeutic abortion, immunogenicity assessments will be done on blood samples obtained after the termination of the pregnancy.

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 48 (Estimated)
Dates: Start 2016-08 (Actual); Primary Completion 2017-11 (Actual); Study Completion 2017-11 (Actual)

PRIMARY OUTCOMES:
Frequency of TV005 and rDEN3Δ30-related adverse events (AEs) | Measured through Day 360
  As classified by both severity and seriousness, through active and passive surveillance
Frequency of viremia | Measured through Day 360

CONTACTS AND LOCATIONS:
Overall Officials: Anna Durbin, MD, Principal Investigator — Center for Immunization Research (CIR), Johns Hopkins School of Public Health
Locations (2):
- United States (2):
  - Center for Immunization Research, Johns Hopkins School of Public Health, Baltimore, Maryland
  - University of Vermont Testing Center, Burlington, Vermont

REFERENCES:
- [Derived] Pierce KK, Durbin AP, Walsh MR, Carmolli M, Sabundayo BP, Dickson DM, Diehl SA, Whitehead SS, Kirkpatrick BD. TV005 dengue vaccine protects against dengue serotypes 2 and 3 in two controlled human infection studies. J Clin Invest. 2024 Feb 1;134(3):e173328. doi: 10.1172/JCI173328. PMID 37971871